CLINICAL TRIAL: NCT02948140
Title: Evaluation of New Diagnostic Methods of Cardio-embolic Related (Atrial Fibrillation) Cerebral Infarction
Acronym: IRMA2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/02; 2016-A00020-51 (Other: ANSM)
Record Dates: First submitted 2016-10-18; First posted 2016-10-28 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: Subdiaphragmatic infarction
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stroke (Experimental)
  Interventions: Procedure: MRI; Procedure: Abdominal scanner

INTERVENTIONS:
Procedure: MRI
Procedure: Abdominal scanner

SUMMARY:
The aim of the study is to estimate the contribution of abdominal imaging by magnetic resonance Imaging (MRI) and abdominal scanner in the detection of subdiaphragmatic infarction associated to the atrial fibrillation in the cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18
* Patient having a CHADS-VAsc Score ≥ 2;
* Patient hospitalized for a secondary established ischemic accident in an atrial fibrillation not anticoagulated (INR<2 and/or receiving antiplatelet (aspirin, clopidogrel)) for less than 14 days;
* Patient affiliated to a national insurance scheme or beneficiary
* Patient having given a written consent

Exclusion Criteria:

* Patient presenting cognitive disorders incompatible with the planned examinations (MRI / SCANNER).
* Pacemaker or implantable defibrillator, or other contraindication in the MRI (metallic eye brightness, intra cerebral clip).
* Contraindication in injected scanner.
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with subdiaphragmatic infarctions detected by abdominal MRI | 14 days

SECONDARY OUTCOMES:
Number of patients with subdiaphragmatic infarctions detected by abdominal scanner | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lapergue, MD, Principal Investigator — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slaoui T, Klein IF, Guidoux C, Cabrejo L, Meseguer E, Abboud H, Lavalllee PC, Mazighi M, Labreuche J, Amarenco P. Prevalence of subdiaphragmatic visceral infarction in cardioembolic stroke. Neurology. 2010 Mar 30;74(13):1030-2. doi: 10.1212/WNL.0b013e3181d76aaa. Epub 2010 Mar 3. PMID 20200339
- [Background] Abboud H, Labreuche J, Gongora-Riverra F, Jaramillo A, Duyckaerts C, Steg PG, Hauw JJ, Amarenco P. Prevalence and determinants of subdiaphragmatic visceral infarction in patients with fatal stroke. Stroke. 2007 May;38(5):1442-6. doi: 10.1161/STROKEAHA.106.476804. Epub 2007 Mar 22. PMID 17379822
- [Background] Flint AC, Tayal AH. The search for paroxysmal atrial fibrillation in cryptogenic stroke: leave no stone unturned. Neurology. 2013 Apr 23;80(17):1542-3. doi: 10.1212/WNL.0b013e31828f1938. Epub 2013 Mar 27. PMID 23535494
- [Background] White H, Boden-Albala B, Wang C, Elkind MS, Rundek T, Wright CB, Sacco RL. Ischemic stroke subtype incidence among whites, blacks, and Hispanics: the Northern Manhattan Study. Circulation. 2005 Mar 15;111(10):1327-31. doi: 10.1161/01.CIR.0000157736.19739.D0. PMID 15769776